CLINICAL TRIAL: NCT01863511
Title: Primary Mode of Therapy in Acute Decompensated Heart Failure:Comparison Between Usual Care Plus Tolvaptan and Ultrafiltration.
Brief Title: Tolvaptan/Ultrafiltration in the Treatment of Acute Heart Failure
Acronym: TUF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Dr. Eugene Chung, Eugene S. Chung MD, FACC, The Christ Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUF-01
Record Dates: First submitted 2013-05-20; First posted 2013-05-29 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-02

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Treatment options for acute decompensated heart failure; Ultrafiltration; tolvaptan
MeSH Terms: interventions — Sodium Potassium Chloride Symporter Inhibitors; Tolvaptan; Ultrafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- usual care (Active Comparator): IV loop diuretics
  Interventions: Drug: loop diuretic
- Usual care plus tolvaptan (Active Comparator): IV loop diuretic plus Tolvaptan 30 mg orally once daily
  Interventions: Drug: loop diuretic; Drug: tolvaptan
- ultrafiltration (Active Comparator): Volume removal through a brachial line extended length catheter or a quad lumen catheter via the internal jugular vein
  Interventions: Procedure: ultrafiltration

INTERVENTIONS:
Drug: loop diuretic
  Arms: Usual care plus tolvaptan; usual care
Drug: tolvaptan
  Arms: Usual care plus tolvaptan
Procedure: ultrafiltration
  Arms: ultrafiltration

SUMMARY:
For patients hospitalized with acute decompensated heart failure,volume removal remains the primary therapeutic objective. The current standard of care remains loop diuretics.The high likelihood of readmissions and poor outcomes highlights the need to examine and improve in-hospital protocols for these patients. Ultrafiltration allows for greater volume removal, less neurohormonal stimulation and greater sodium removal.However it is associated with increased costs, line complications, and relative immobility during treatment. Tolvaptan in addition to diuretic therapy has been shown to improve the amount of volume removed compared to diuretic alone.

The study proposes to compare the strategy of adding tolvaptan to usual care with ultrafiltration as primary mode of therapy in acute decompensated HF(ADHF) patients.

Hypothesis: addition of tolvaptan to usual care for hospitalized HF patients will result in:

* greater volume and weight reduction compared with usual care
* similar efficacy outcomes compared with ultrafiltration, with less complications of therapy

DETAILED DESCRIPTION:
Study design is a prospective randomized open labeled and unblinded comparison of two different approaches to volume removal. Enrolled patients will be evaluated for target weight to be removed. Patients will be randomized to usual care (UC), usual care plus tolvaptan (UC+T) or ultrafiltration (UF), within 12 hours of presentation.

Treatment in the UC and UC+T arms will begin with a furosemide bolus(double the home dose or if unavailable, 60mg) and continue with a drip(10 or 20 mg/hr). In addition the UC+T group will be treated with tolvaptan 30 mg orally once daily.

Patients in the UF arm will be treated with UF administered through a brachial line or a catheter in the internal jugular vein. Loop and thiazide diuretics will be discontinued, although aldosterole antagonists will be continued.

Urinary neutrophil gelatinase associated lipocalcin(uNGAL)levels are elevated in renal dysfunction and may be a sensitive biomarker to distinguish between intrinsic renal damage and reversible, transient prerenal azotemia.Characterizing the changes in uNGAL levels during the course of ADHF therapy, in comparison with patient weight, BUN and creatinine levels is an important step in establishing the role of this potential promising biomarker in ADHF treatment strategies.

Protocol highlights for all patients include:

Baseline labs and daily through day 4 and at discharge(BMP, BNP, CBC, urine creatinine and sodium, uNGAL)

* Daily am weights
* Daily volume status:total intake, urine output, ultrafiltrate volume
* Collect all urine and ultrafiltrate in a 24 hour collection bag, record volume, creatinine and Na levels
* length of stay
* hospital day 4: Minnesota Living with Heart Failure questionnaire
* Cost of hospitalization

ELIGIBILITY:
Inclusion Criteria:

* 2 of 3 physical exam findings of volume overload (rales, JVP over 5 cm and edema)
* BNP over 300
* no contraindication to ultrafiltration (line insertion, heparin use)

Exclusion Criteria:

* serum creatinine > 3mg/dL or Na > 145
* inotrope or vasopressor dependency
* active infection, including urinary tract
* resynchronization therapy or coronary intervention in past 30 days
* life expectancy less than 6 months
* hypertrophic obstructive cardiomyopathy with peak resting gradient > 20 mmHg
* IV contrast or NSAID use in the past 1 week (uNGAL related requirement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Net change in weight | day 1,2,3,4,5

SECONDARY OUTCOMES:
net volume loss | day 1,2,3,4,5
urinary NGAL | Day 1,2,3,4,5
dyspnea score | baseline and day 5
BNP change from admission to discharge | baseline and day 5
serum creatinine change | Day 1,2,3,4,5
serum sodium and potassium changes | baseline through day 5
Quality of Life | day 4 of hospital stay
all cause readmission | 30 day
all cause death | 30 day

OTHER OUTCOMES:
nursing intensity | day 1,2,3,4,5
peripheral vs. central access, number of filters used, complications of heparin use | day 1,2,3,4,5

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S Chung, MD, Principal Investigator — The Christ Hospital
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Srivastava M, Harrison N, Caetano AFS, Tan AR, Law M. Ultrafiltration for acute heart failure. Cochrane Database Syst Rev. 2022 Jan 21;1(1):CD013593. doi: 10.1002/14651858.CD013593.pub2. PMID 35061249